CLINICAL TRIAL: NCT00479141
Title: A Cluster-Randomized Trail to Evaluate the Efficacy of a Combined Individual- and Community-Based Behavioral Intervention to Improve Quality of Life (QOL) For HIV-Positive Villagers in Rural China
Brief Title: A Cluster-Randomized Intervention Trial to Improve Quality of Life for HIV-Infected Individuals in Anhui, China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CIPRA CH 002B
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Treatment Experienced; Complementary Therapies
MeSH Terms: conditions — HIV Infections

ARMS (2):
- 1 (Experimental): HIV infected participants and their families
  Interventions: Behavioral: HIV skills training
- 2 (Experimental): Popular Opinion Leaders (POL) participants
  Interventions: Behavioral: Popular Opinion Leaders training

INTERVENTIONS:
Behavioral: HIV skills training — Eight 2-hour group skills training sessions will occur during Weeks 1 through 8 and booster sessions will occur every two months during Months 3 through 15
  Arms: 1
Behavioral: Popular Opinion Leaders training — Two-hour training sessions about anti-stigma and anti-discrimination will occur for 4 weeks, followed by support meetings every 2 months during Months 2 through 13.
  Arms: 2

SUMMARY:
The HIV epidemic in China has reached a phase of exponential growth; the number of new infections has been steadily increasing over the past decade. The purpose of this study is to evaluate the effectiveness of a Combined Individual- and Community-Based Behavioral Intervention to Improve Quality of Life for HIV-Positive Villagers and decrease HIV related stigma in Rural China.

DETAILED DESCRIPTION:
Over the past decade, the rates of HIV infection and death due to HIV/AIDS have been steadily increasing in China. The China Comprehensive AIDS Response (China CARES) program was developed in 2003 in order to help poor counties and those with severe epidemic problems increase public awareness and improve knowledge about epidemic diseases such as HIV. Currently, behavioral interventions focusing on individual skills training and self-efficacy building for HIV infected individuals are not included in China CARES. Fuyang, Anhui Province, China has a high rate of HIV infected individuals, many of whom were former plasma donors (FPDs) and would benefit from HIV skills training.

In 2004, CIPRA conducted a study (CIPRA CH 002A), entitled "A Qualitative Study for the Development of an Intervention Among HIV-Positive Former Plasma Donors (FPDs) in Fuyang, Anhui Province, China," which provided insight into HIV infected individuals in Fuyang, Anhui Province, China. According to the results of CIRPA CH 002A, most HIV infected individuals described their QOL as poor. The factors affecting their poor QOL include poverty, poor health, stigma and discrimination. Participants in the CIPRA CH 002A study showed interest in learning more about HIV/AIDS disease and treatment. This study will last 18 months. HIV infected participants and their families will attend eight 2-hour group skills training sessions during Weeks 1 through 8, and booster sessions every two months during Months 3 through 15. Popular Opinion Leaders (POL) participants will attend 4 weeks of 2-hour training sessions about anti-stigma and anti-discrimination, followed by support meetings every 2 months during Months 2 through 13. Some participants will complete cross-sectional surveys evaluating the levels of stigma and discrimination in the community at study entry and at Months 6 and 12 following completion of POL training. All participants will complete follow-up visits at Months 6 and 12.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Individuals:

* HIV infected
* Resident of Funan County or Yingzhou District, Anhui Province, China
* Willing to provide location information

Inclusion Criteria for Family members of HIV Infected Individuals:

* Resident of Funan County or Yingzhou District, Anhui Province, China
* Family member of HIV infected participant

Inclusion Criteria for POLs:

* Identified as an influential member of the community
* Resident of Funan County or Yingzhou District, Anhui Province, China
* Willing to attend training and follow-up meetings Note: Both HIV infected and non HIV infected individuals may participate as POLs

Inclusion Criteria for Cross-Sectional Survey Participants:

* Resident of Funan County or Yingzhou District, Anhui Province, China
* Randomly selected and invited to participate in study

Exclusion Criteria for HIV Infected Individuals:

* Spent more than 6 months outside the community within the year prior to study entry
* Permanent disability (e.g., deafness, serious mental illness, mental retardation)
* Has not made contact with study staff after three attempts

Exclusion Criteria for Family Members of HIV Infected Individuals:

* Permanent disability (e.g., deafness, serious mental illness, mental retardation)

Exclusion Criteria for POLs:

* Spent more than 6 months outside the community within the year prior to study entry
* Permanent disability (e.g., deafness, serious mental illness, mental retardation)

Exclusion Criteria for Cross-Sectional Survey Participants:

* Spent more than 6 months outside the community within the year prior to study entry
* Permanent disability (e.g., deafness, serious mental illness, mental retardation)
* Has not made contact with study staff after three attempts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3199 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study HIV Health Survey (MOS-HIV) score in HIV infected participants | Throughout study

SECONDARY OUTCOMES:
Level of stigma among community members, including HIV knowledge | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, MD, PhD, Study Chair — Division of Health Education and Behavioral Intervention, National Center for AIDS/STD Control and Prevention, Chinese Center for Disease Control and Prevention; Jie Xu, MD, MS, MPH, Study Chair — Division of Health Education and Behavioral Intervention, National Center for AIDS/STD Control and Prevention, Chinese Center for Disease Control and Prevention
Locations (1):
- Fuyang CDC Office, Beijing, China

REFERENCES:
- [Background] Wu Z, Sullivan SG, Wang Y, Rotheram-Borus MJ, Detels R. Evolution of China's response to HIV/AIDS. Lancet. 2007 Feb 24;369(9562):679-90. doi: 10.1016/S0140-6736(07)60315-8. PMID 17321313
- See also: Click here for more information about CIPRA CH 002A: HIV Assessment in Fuyang, Anhui Province, China — http://clinicaltrials.gov/show/NCT00094354